CLINICAL TRIAL: NCT03108664
Title: HELIX, a Double-masked Study of SYL1001 in Patients With Moderate to Severe Dry Eye
Brief Title: HELIX, a Double-masked Study of SYL1001 in Patients With Moderate to Severe Dry Eye Disease (DED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sylentis, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYL1001_IV; 2016-003903-79 (EudraCT Number)
Record Dates: First submitted 2017-03-30; First posted 2017-04-11 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-09

CONDITIONS: Dry Eye Disease
Keywords: SYL1001; siRNA
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 11.25 mg/mL SYL1001 ophthalmic solution (Experimental): 1 drop of 11.25 mg/mL SYL1001 ophthalmic solution in the affected eye(s) q.d
  Interventions: Drug: SYL1001 ophthalmic solution
- Vehicle ophthalmic solution (Experimental): 1 drop of vehicle ophthalmic solution in the affected eye(s) q.d
  Interventions: Drug: Vehicle opthalmic solution

INTERVENTIONS:
Drug: SYL1001 ophthalmic solution — 1 drop in the affected eye
  Arms: 11.25 mg/mL SYL1001 ophthalmic solution
Drug: Vehicle opthalmic solution — 1 drop in the affected eye
  Arms: Vehicle ophthalmic solution

SUMMARY:
The purpose of this study is to determine whether SYL1001 ophthalmic solution is safe and effective in the treatment of signs and symptoms of Dry Eye Disease.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* ≥ 18 years old
* Give written informed consent to participate in the study after having been informed of the study design, objectives and possible derived risks
* Common symptoms of persistent, daily, moderate to severe dry eye lasting more than six months.
* Use of artificial tears
* VAS scale for eye discomfort/pain between 30 - 80
* CFS ≥ 2 and ≤ 4 on the Oxford scale
* TBUT < 10 seconds
* Hyperemia score ≥ 1 (McMonnies scale)
* Schirmer's test without anesthesia ≥ 2 and < 10 mm/5min in the eye
* Corrected visual acuity ≥ 0.7 logMAR

Exclusion Criteria:

* Pregnant or breastfeeding females or those with a positive pregnancy test.
* Females of childbearing potential who will not use a medically acceptable contraceptive method from selection and during the whole study.
* Current relevant disease, including respiratory disease, cardiovascular, endocrine, neurological, haematological, renal, neoplasic, hepatopathy, gastrointestinal distress, hypertension, or infectious acute processes.
* Past history of a chronic o recurring condition that could interfere with study according to the investigator's judgement.
* Concomitant use of other drugs with analgesic activity by any route of administration at the enrolment period.
* Changes in any ocular and/or systemic concomitant medication one month prior to the study commencement and during the study development.
* Changes on the preestablished artificial tears dosage 15 days prior to the study commencement and during the study development.
* Cyclosporine treatment initiation or changes in cyclosporine dosage or dosing regimen during the 6 months prior to enrolment.
* Previous history of drug hypersensitivity.
* Use of contact lenses
* Case history of drug or alcohol abuse or dependence.
* Relevant abnormal laboratory results as judged by the investigator
* Previous refractive surgery
* Participation in a clinical trial within 2 months before the enrolment visit
* Relevant ocular pathology judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Visual Analogue Scale (VAS) scores for eye discomfort/pain as a measurement of SYL1001 effect versus vehicle | 28 days
Change from baseline in Corneal Fluorescein Staining (CFS) total scores obtained on the Oxford scale as a measurement of SYL1001 effect versus vehicle | 28 days
Change from baseline in conjunctival hyperaemia scores based on the McMonnies scale as a measurement of SYL1001 effect versus vehicle | 28 days

SECONDARY OUTCOMES:
Assessment of Adverse Events Appearance as a measure of SYL1001 tolerability | 28 days

CONTACTS AND LOCATIONS:
Locations (40):
- Estonia (3):
  - East Tallin Central Hospital, Tallinn
  - Eye Clinic Dr. Krista Turman, Tallinn
  - Tartu University Hospital, Tartu
- Germany (8):
  - Augenzentrum Nord-West, Ahaus
  - Uniklinik Köln Zentrum für Augenheilkunde, Cologne
  - Universitäts-Augenklinik Düsseldorf, Düsseldorf
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum des Saarlandes, Homburg
  - Klinik für Augenheilkunde Universitätsklinikum Schleswig-Holstein, Kiel
  - Universitätsklinikum Leipzig AöR Klinik und Poliklinik für Augenheilkunde, Leipzig
  - Augenklinik der Ludwig-Maximilian Universität München, München
- Italy (4):
  - AOU Careggi, Florence
  - Ospedale San Giuseppe, Milan
  - Farmacia Azienda Ospedaliera di Padova, Padua
  - A.O.U. Pisana, Pisa
- Portugal (3):
  - Hospital de Braga, Braga
  - Centro Hospitalar e Universitário de Coimbra, Coimbra
  - Hospital Lusiadas Lisboa, Lisbon
- Slovakia (7):
  - Bellet s.r.o, Martin
  - Optomedic s.r.o, Štúrovo
  - Oftalmologická ambulancia, Trenčín
  - Fakultná nemocnica Trenčín,, Trenčín
  - OPHTHAMED, s.r.o.,, Žilina
  - VIKOM s.r.o, Žilina
  - Fakultná nemocnica s poliklinikou Žilina, Žilina
- Spain (15):
  - Hospital Universitario Príncipe de Asturias, Alcalá de Henares, Madrid
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Instituto Oftalmológico Fernández Vega, Oviedo, Principality of Asturias
  - Institut Català de la Retina, Barcelona
  - Instituto de Oftalmología del Hospital Clínic de Barcelona Casa de la Maternitat, Barcelona
  - Instituto de Microcirugía Ocular (IMO), Barcelona
  - Centro de Oftalmología Barraquer, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario la Paz, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - FISABIO Oftalmología Médica (FOM), Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Provincial Nuestra Señora de Gracia, Zaragoza